CLINICAL TRIAL: NCT07256301
Title: A Multicenter, Open-Label, Phase Ib Clinical Trial to Evaluate the Safety, Pharmacokinetic, and Pharmacodynamic Profiles of Multiple Doses of the Humanized Monoclonal Antibody EA5 in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: A Phase Ib, Multicenter, Open-Label Study of Multiple-Dose EA5 in Adults With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Lanyi Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C-EA5-2401
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: PNH - Paroxysmal Nocturnal Hemoglobinuria
Keywords: EA5、PNH、Paroxysmal Nocturnal Hemoglobinuria、C5 complement inhibitor
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 and Cohort 1' (Experimental): Participants were administered EA5 900 milligram (mg) on Day 1 and Day 8, EA5 900 mg on Day 15, and then EA5 900 mg every 4 weeks for 2 doses.
  Interventions: Biological: EA5
- Cohort 2 and Cohort 2' (Experimental): Participants were administered EA5 900 milligram (mg) on Day 1 and Day 8, EA5 1200 mg on Day 15, and then EA5 1200 mg every 4 weeks for 2 doses.
  Interventions: Biological: EA5
- Cohort 3 (Experimental): Participants were administered EA5 900 milligram (mg) on Day 1 and Day 8, EA5 1400 mg on Day 15, and then EA5 1400 mg every 4 weeks for 2 doses.
  Interventions: Biological: EA5

INTERVENTIONS:
Biological: EA5 — All treatments were given as IV infusions.

SUMMARY:
This is a multicenter, open-label, Phase Ib clinical trial designed to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple doses of the humanized monoclonal antibody EA5 in adult patients with paroxysmal nocturnal hemoglobinuria (PNH).

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase Ib clinical trial designed to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple doses of the humanized monoclonal antibody EA5 in adult patients with paroxysmal nocturnal hemoglobinuria (PNH). The study plans to enroll 24-26 PNH patients. The primary objective is to assess the incidence and severity of adverse events (AEs) from baseline to Week 14.The treatment period is divided into a Loading Phase (Day 1 to Day 14) and a Maintenance Phase (Day 15 to Day 85). During the maintenance phase, patients will be assigned to one of three dose cohorts: Cohort 1/Cohort 1' (900 mg, IV, Q4W), Cohort 2/Cohort 2' (1200 mg, IV, Q4W), and Cohort 3 (1400 mg, IV, Q4W). Cohorts 1-3 are for patients previously naive to complement inhibitor therapy, while Cohorts 1'-2' are for patients recently naive to complement inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years.
* Body weight between 40 kg and 100 kg (inclusive) at screening.
* Patients diagnosed with PNH, confirmed by flow cytometry demonstrating a PNH clone size (glycosylphosphatidylinositol-anchored protein-deficient granulocytes or monocytes) of ≥10% in peripheral blood, and meeting one of the following criteria:

  * a) Previously naive to complement inhibitor therapy; or
  * b) Previously treated with a complement inhibitor, which has been discontinued for ≥5 half-lives prior to screening.
* Lactate dehydrogenase (LDH) level ≥1.5 times the upper limit of normal (ULN) at screening.
* Presence of one or more of the following PNH-related signs or symptoms within 3 months prior to screening: fatigue, hemoglobinuria, abdominal pain, shortness of breath (dyspnea), anemia (hemoglobin <10 g/dL), history of major thrombotic event (including thrombosis), dysphagia, or erectile dysfunction; or a history of packed red blood cell (pRBC) transfusion due to PNH.
* Vaccination against Neisseria meningitidis(serogroups A, C, W, Y) within <3 years prior to the initiation of study treatment; OR if not previously vaccinated, receipt of the meningococcal vaccine (MPV-ACYW) at least 14 days prior to the first dose of the investigational product. If the vaccine is administered within 14 days before dosing, antibiotic prophylaxis must be provided until 2 weeks post-vaccination.
* Vaccination against Streptococcus pneumoniaeaccording to national vaccination recommendations (e.g., ACIP guidelines). OR if not previously vaccinated, receipt of the pneumococcal vaccine at least 14 days prior to the first dose of the investigational product. If the vaccine is administered within 14 days before dosing, antibiotic prophylaxis must be provided until 2 weeks post-vaccination.
* For patients receiving concomitant therapies (e.g., immunosuppressants, corticosteroids, iron supplements, anticoagulants, erythropoiesis-stimulating agents): the dose must have been stable for ≥28 days prior to the first dose of the investigational product.
* Platelet count ≥30 × 10^9/L at screening (without transfusion support within 7 days), and absolute neutrophil count (ANC) ≥0.5 × 10^9/L (without short-acting granulocyte colony-stimulating factor (G-CSF) within 14 days or long-acting G-CSF within 28 days).
* Adequate liver function, defined as alanine aminotransferase (ALT) ≤3 × ULN, OR both direct bilirubin and alkaline phosphatase (ALP) ≤2 × ULN at screening.
* Adequate renal function, defined as serum creatinine ≤2.5 × ULN and an estimated creatinine clearance ≥30 mL/min as calculated by the Cockcroft-Gault formula.
* Male subjects must agree to use effective contraception (including vasectomy, abstinence, or condom) from screening until 6 months after the final study intervention. Women of childbearing potential (WOCBP) must have a negative blood pregnancy test at screening and baseline. During the study and for 6 months thereafter, all subjects and their partners must agree to use effective contraceptive measures (Note: contraceptive measures include both pharmacological and non-pharmacological methods).
* Ability to understand the procedures and methods of the study, willingness to provide written informed consent, and commitment to strictly adhere to the clinical study protocol to complete the study.

Exclusion Criteria:

* History of allogeneic bone marrow transplantation.
* History of Neisseria meningitidisinfection within 6 months prior to screening and before the first dose.
* Known or suspected immunodeficiency (e.g., history of frequent or recurrent infections).
* Known or suspected hereditary complement deficiency.
* Evidence of active tuberculosis (TB) within 6 months prior to screening, or a history of active TB without having completed an appropriate, documented course of treatment; OR chest X-ray (posteroanterior and lateral) or CT scan findings during the 3 months prior to screening or during the screening period that suggest the presence of active TB infection.
* History of major surgery (Grade 3 or 4 surgery) within 3 months prior to the first dose.
* Presence of an autoimmune disease, OR use of systemic immunosuppressive/immunomodulatory agents (including, but not limited to, methotrexate, cyclosporine, mycophenolate, tacrolimus, penicillamine, sulfasalazine, hydroxychloroquine, azathioprine, cyclophosphamide) for the treatment of inflammatory diseases within 12 weeks or 5 half-lives (whichever is longer) prior to screening.
* Active systemic bacterial, viral, or fungal infection within 14 days prior to the first dose; OR requirement for hospitalization or intravenous antibiotic therapy for an infection between 28 days prior to screening and the first dose; OR requirement for oral antibiotic therapy for an infection between 14 days prior to screening and the first dose.
* Occurrence of fever (≥38°C) within 7 days prior to the first drug administration.
* Administration of any live-attenuated vaccine within 1 month prior to the first dose.
* History of malignancy within 5 years prior to screening and before the first dose, with the following exceptions: patients with any malignancy that has been treated with curative intent and who have been disease-free and off treatment for >5 years prior to the first dose may be enrolled. Patients with a history of basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situof the cervix that has been cured with no evidence of recurrence at any time prior to the first dose may be enrolled. Patients with a history of low-grade, early-stage prostate cancer (Gleason score ≤6, Stage 1 or 2) not requiring treatment at any time prior to the first dose may be enrolled.
* History of allergy to any component of EA5, including a history of hypersensitivity to human, humanized, or murine monoclonal antibodies, or known hypersensitivity to any excipient of the product.
* Any contraindication to receiving the meningococcal vaccination and/or antibiotic prophylaxis (e.g., beta-lactam antibiotics, ciprofloxacin) as required by the study protocol.
* Participation in another interventional therapeutic clinical trial involving an investigational drug or receipt of any experimental therapy within 3 months (or within 5 half-lives of the investigational agent, whichever is longer) prior to screening.
* History of drug abuse within 12 months prior to screening, as judged by the investigator.
* Alcohol abuse, or regular alcohol consumption exceeding 14 units per week within 6 months prior to screening (1 unit of alcohol ≈ 360 mL of beer, or 45 mL of 40% spirits, or 150 mL of wine).
* Splenectomy performed within ≤6 months prior to screening.
* Positive for hepatitis C virus (HCV) antibody at screening (except for those with a negative HCV RNA result), positive for human immunodeficiency virus (HIV) antibody, positive for anti-Treponema pallidumantibody (TP-Ab) (except for those with a negative RPR or TRUST test), OR positive for hepatitis B virus (HBV) surface antigen (HBsAg) (except for those with an HBV DNA level ≤1000 IU/mL).
* History of or ongoing cryoglobulinemia at the time of screening.
* History of myelodysplastic syndromes (MDS), with a Revised International Prognostic Scoring System (IPSS-R) risk category of Intermediate, High, or Very High.
* Any other condition that, in the opinion of the investigator, renders the subject unsuitable for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Baseline up to Week 14
  TEAEs were defined as AEs that occurred on or after the date and time of study drug administration, or those that first occurred before dosing but worsened in frequency or severity after study drug administration. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of EA5 | Baseline up to Week 14
  Blood samples were collected for analysis of Cmax
Time To Maximum Observed Serum Concentration (Tmax) of EA5 | Baseline up to Week 14
  Blood samples were collected for analysis of Tmax
Area Under The Serum Concentration Versus Time Curve From Time Zero To The Time of The Last Quantifiable Concentration (AUC0-t) of EA5 | Baseline up to Week 14
  Blood samples were collected for analysis of AUC0-t
Area Under The Serum Concentration Versus Time Curve From Time Zero (Dosing) To Infinity (AUCinf) of EA5 | Baseline up to Week 14
  Blood samples were collected for analysis of AUCinf
Terminal Elimination Rate Constant (λz) of Serum EA5 | Baseline up to Week 14
  Blood samples were collected for analysis of λz
Terminal Elimination Half-life (t½) of Serum EA5 | Baseline up to Week 14
  Blood samples were collected for analysis of t½
Total Clearance (CL) of EA5 | Baseline up to Week 14
  Blood samples were collected for analysis of CL
Percent Change From Baseline in Free Complement Component 5 (C5) | Baseline up to Week 14
  Blood samples were collected for analysis of free C5 concentrations.
Percent Change From Baseline in Total Complement C5 | Baseline up to Week 14
  Blood samples were collected for analysis of total C5 concentrations.
Percent Change From Baseline in determination of terminal complement activity in serum | Baseline up to Week 14
  Blood samples were collected for analysis of determination of terminal complement activity
Percentage of Participants With Positive Anti-Drug Antibody (ADA) | Baseline up to Week 14
  Blood samples were collected to evaluate antibody response through development of ADAs.

CONTACTS AND LOCATIONS:
Overall Officials: Fengkui Zhang, Dr., Principal Investigator — The Institute of Hematology & Blood Diseases Hospital (Chinese Academy of Medical Sciences); Hongyan Tong, Dr., Principal Investigator — The First Affiliated Hospital, Zhejiang University School of Medicine, Chengzhan Campus
Locations (2):
- China (2):
  - The Institute of Hematology & Blood Diseases Hospital (Chinese Academy of Medical Sciences), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Chengzhan Campus, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided